CLINICAL TRIAL: NCT04770350
Title: Open Label Study for the Use of Transcranial Ultrasound for Treatment of Age-Related Frailty
Acronym: fUS-ARF
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Neurological Associates of West Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: fUS-Frailty
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Frailty; Aging
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Experimental (Experimental): Participants will undergo ten to thirty minutes of transcranial ultrasound treatment. The sanitation device will be aimed at the hypothalamus. Targeting will include reference to scalp fiducials based on the obtained MRI; confirmation of target accuracy will either be obtained by Doppler waveform confirmation or optical tracking technology which co-registers patient neuroimaging with real space.
  Interventions: Device: Focused Ultrasound

INTERVENTIONS:
Device: Focused Ultrasound — The DWL Doppler ultrasound device enables visual and auditory waveform confirmation of the middle cerebral artery, and optical tracking technology (e.g., AntNeuro Visor2™ system) may be used in tandem with the Brainsonix ultrasound device to track a patient's brain in virtual space as well as their physical location, thereby ensuring accurate placement.

SUMMARY:
The purpose of this Phase I open label study is to evaluate longer term tolerability and potential effectiveness of transcranial ultrasound in people with age-related frailty.

DETAILED DESCRIPTION:
This study is designed to evaluate the safety and efficacy of focused ultrasound in patients with age-related frailty characterized by reduced physical and immunological functioning. The safety of this protocol will be closely monitored and data will be used to determine whether any significant safety issues exist when using focused ultrasound. Adverse events will be noted whenever they occur but will be recorded at the time of the procedure and throughout routine follow-ups, which will persist weekly throughout the duration of the active study protocol. Patients deemed potentially appropriate candidates for focused ultrasound therapy will be treated with 8 sessions of transcranial ultrasound, each of which consists of 10 to 30 minutes of active administration. Clinical and safety outcome measures will be obtained throughout and after completion of the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age eligibility requirements fall in a range from 60 to 95 years of age
* Clinical appraisal by physician indicating signs of frailty (apart from a co-occuring condition), scoring 3<x<7 as denoted by the CSHA Clinical Frailty Scale (Rockwood, Song, MacKnight, et al, 2005; Golpanian, DiFede, Pujol, et al., 2016)
* MRI of the brain including volume measurement of the hypothalamus

Exclusion Criteria:

* Subjects unable to give informed consent
* Subjects who would not be able to lay down without excessive movement in a calm environment sufficiently long enough to be able to achieve sleep
* Pregnancy, women who may become pregnant or are breastfeeding
* Advanced terminal illness
* Subjects with scalp rash or open wounds on the scalp (for example from treatment of squamous cell cancer)

Ages: 45 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Frailty Scale (CFS) | Baseline
  The CFS is a 9-point scoring guide for physicians to use upon clinical appraisal of frailty-related symptoms. The lowest rating is 1 ("Very Fit") and the highest rating is 9 ("Terminally Ill"). The range of acceptable ratings for screened participants is from 3 ("Managing Well") to 7 ("Severely Frail").
Clinical Frailty Scale (CFS) | Final Evaluation (8 weeks from baseline)
  The CFS is a 9-point scoring guide for physicians to use upon clinical appraisal of frailty-related symptoms. The lowest rating is 1 ("Very Fit") and the highest rating is 9 ("Terminally Ill"). The range of acceptable ratings for screened participants is from 3 ("Managing Well") to 7 ("Severely Frail"). Scoring on the CFS will be noted as significant for those who improve by at least one level.

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB) | Baseline
  The SPPB is a series of tests used to evaluate lower extremity function and mobility in older people. The test consists of three major components, each of which are scored independently: 3 static balance tests, gait speed, and five timed sit-to-stand tests. Points are assigned based on performance, with a maximum possible score of 12 points. Higher scores are indicative of better functioning. A score of 0 on any item indicates lack of ability or functioning. The minimum clinically important difference for the total SPPB score is 1 point.
Short Physical Performance Battery (SPPB) | Final Evaluation (8 weeks from baseline)
  The SPPB is a series of tests used to evaluate lower extremity function and mobility in older people. The test consists of three major components, each of which are scored independently: 3 static balance tests, gait speed, and five timed sit-to-stand tests. Points are assigned based on performance, with a maximum possible score of 12 points. Higher scores are indicative of better functioning. A score of 0 on any item indicates lack of ability or functioning. The minimum clinically important difference for the total SPPB score is 1 point.
Multidimensional Fatigue Inventory (MFI) | Baseline
  The MFI is a 20-item scale designed to evaluate five dimensions of fatigue: general fatigue, physical fatigue, reduced motivation, reduced activity, and mental fatigue. Respondents use a scale ranging from 1 to 7 to indicate how aptly certain statements regarding fatigue represent their experiences. Several positively phrased items are reverse- scored. Higher total scores correspond with more acute levels of fatigue. Responses for the Multidimensional Fatigue Inventory will be defined as clinically significant when there is a 2-point difference.
Multidimensional Fatigue Inventory (MFI) | Final Evaluation (8 weeks from baseline)
  The MFI is a 20-item scale designed to evaluate five dimensions of fatigue: general fatigue, physical fatigue, reduced motivation, reduced activity, and mental fatigue. Respondents use a scale ranging from 1 to 7 to indicate how aptly certain statements regarding fatigue represent their experiences. Several positively phrased items are reverse- scored. Higher total scores correspond with more acute levels of fatigue. Responses for the Multidimensional Fatigue Inventory will be defined as clinically significant when there is a 2-point difference.
Montreal Cognitive Assessment (MoCA) | Baseline
  The MoCA evaluates frontal-executive functions (e.g., verbal abstraction and mental calculation), language (e.g., confrontation naming, phonemic fluency), orientation (e.g., person, place, date, day of the week, and time), visuospatial construction (e.g., simple figure copy), divided visual attention, and immediate and delayed memory of unstructured information. MoCA scores range from 0-30 possible points; 26 or greater is considered to reflect normal cognitive status.
Montreal Cognitive Assessment (MoCA) | Final Evaluation (8 weeks from baseline)
  The MoCA evaluates frontal-executive functions (e.g., verbal abstraction and mental calculation), language (e.g., confrontation naming, phonemic fluency), orientation (e.g., person, place, date, day of the week, and time), visuospatial construction (e.g., simple figure copy), divided visual attention, and immediate and delayed memory of unstructured information. MoCA scores range from 0-30 possible points; 26 or greater is considered to reflect normal cognitive status.
Beck Depression Inventory (BDI-II) | Baseline
  The BDI-II is a 21-question multiple-choice self-report inventory. Each question involves four possible responses, ranging in intensity from "0" (this item does not apply) to "3" (this item applies severely). The test is scored as the sum of all of the response values; this number is used to determine the severity of depressive symptoms. A score of 0 to 3 is possible for each question with a maximum total score of 63 points. The standard cutoff scores are as follows: 0-13 total points = minimal depression; 14-19 total points = mild depression; 20-28 total points = moderate depression; and 29-63 total points = severe depression. A reduction in the total score by at least 30% is considered to be clinically significant.
Beck Depression Inventory (BDI-II) | Final Evaluation (8 weeks from baseline)
  The BDI-II is a 21-question multiple-choice self-report inventory. Each question involves four possible responses, ranging in intensity from "0" (this item does not apply) to "3" (this item applies severely). The test is scored as the sum of all of the response values; this number is used to determine the severity of depressive symptoms. A score of 0 to 3 is possible for each question with a maximum total score of 63 points. The standard cutoff scores are as follows: 0-13 total points = minimal depression; 14-19 total points = mild depression; 20-28 total points = moderate depression; and 29-63 total points = severe depression. A reduction in the total score by at least 30% is considered to be clinically significant.
Beck Anxiety Inventory (BAI) | Baseline
  The BAI is a 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety symptoms. Each of the 21 items asks whether the patient has experienced various anxiety symptoms in the last two weeks, and if so, how severely. Each question/answer is scored on a scale value of "0" (not at all) to "3" (severely). Higher total scores indicate more severe anxiety symptoms. The maximum total score possible is 63 points. The standard cutoff scores are: 0-7 = minimal anxiety; 8-15 = mild anxiety; 16-25 = moderate anxiety; 26-63 = severe anxiety. A reduction in score by at least 30% is considered clinically meaningful.
Beck Anxiety Inventory (BAI) | Final Evaluation (8 weeks from baseline)
  The BAI is a 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety symptoms. Each of the 21 items asks whether the patient has experienced various anxiety symptoms in the last two weeks, and if so, how severely. Each question/answer is scored on a scale value of "0" (not at all) to "3" (severely). Higher total scores indicate more severe anxiety symptoms. The maximum total score possible is 63 points. The standard cutoff scores are: 0-7 = minimal anxiety; 8-15 = mild anxiety; 16-25 = moderate anxiety; 26-63 = severe anxiety. A reduction in score by at least 30% is considered clinically meaningful.
Community Healthy Activities Model Program for Seniors (CHAMPS) | Baseline
  This self-report questionnaire assesses weekly frequency and duration of a variety of lifestyle physical activities that are meaningful and appropriate for older adults. It includes activities of various intensities (from light to vigorous) such as walking, running, hiking, swimming, bicycling, dancing, tennis, aerobics, yoga/tai chi, gardening, and housework. Intensity is reflected in the item stem (e.g., light and heavy gardening are separate items). The questionnaire is self-administered, although it can be interviewer administered. It is formatted to accommodate increasing visual problems with age by using a large font, adequate space on the page, and high contrast. A total caloric expenditure is calculated based on reported participant activity. Responses for the CHAMPS questionnaire will be defined as clinically significant when there is a 8 kcal/kg/week difference.
Community Healthy Activities Model Program for Seniors (CHAMPS) | Final Evaluation (8 weeks from baseline)
  This self-report questionnaire assesses weekly frequency and duration of a variety of lifestyle physical activities that are meaningful and appropriate for older adults. It includes activities of various intensities (from light to vigorous) such as walking, running, hiking, swimming, bicycling, dancing, tennis, aerobics, yoga/tai chi, gardening, and housework. Intensity is reflected in the item stem (e.g., light and heavy gardening are separate items). The questionnaire is self-administered, although it can be interviewer administered. It is formatted to accommodate increasing visual problems with age by using a large font, adequate space on the page, and high contrast. A total caloric expenditure is calculated based on reported participant activity. Responses for the CHAMPS questionnaire will be defined as clinically significant when there is a 8 kcal/kg/week difference.
Grip Strength (Dynamometer Performance) | Baseline
  Participants will be asked to demonstrate grip strength in standard fashion for clinical evaluation. Using the JAMAR Technologies Hydraulic Hand Dynamometer, participants will squeeze the instrument with their dominant hand and generate a reading of grip strength in the output reading (units = kg). The MCID of the grip strength test is a change of at least 5.0 kg.
Grip Strength (Dynamometer Performance) | Final Evaluation (8 weeks from baseline)
  Participants will be asked to demonstrate grip strength in standard fashion for clinical evaluation. Using the JAMAR Technologies Hydraulic Hand Dynamometer, participants will squeeze the instrument with their dominant hand and generate a reading of grip strength in the output reading (units = kg). The MCID of the grip strength test is a change of at least 5.0 kg.
Global Rating of Change (GRC) | Final Evaluation (8 weeks from baseline)
  The GRC consists of a single likert-scale ranging from "-5" (very much worse) to "0" (neutral/no change) to "5" (very much better). The GRC is obtained in an interview format to assess a patient's perceived change in status following a treatment. A score that is at least 2 or greater is considered to indicate clinically significant change.

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Jordan, MD, Principal Investigator — Neurological Associates - The Interventional Group
Locations (1):
- Neurological Associates of West Los Angeles, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tompkins BA, DiFede DL, Khan A, Landin AM, Schulman IH, Pujol MV, Heldman AW, Miki R, Goldschmidt-Clermont PJ, Goldstein BJ, Mushtaq M, Levis-Dusseau S, Byrnes JJ, Lowery M, Natsumeda M, Delgado C, Saltzman R, Vidro-Casiano M, Da Fonseca M, Golpanian S, Premer C, Medina A, Valasaki K, Florea V, Anderson E, El-Khorazaty J, Mendizabal A, Green G, Oliva AA, Hare JM. Allogeneic Mesenchymal Stem Cells Ameliorate Aging Frailty: A Phase II Randomized, Double-Blind, Placebo-Controlled Clinical Trial. J Gerontol A Biol Sci Med Sci. 2017 Oct 12;72(11):1513-1522. doi: 10.1093/gerona/glx137. PMID 28977399
- [Background] Zhang Y, Kim MS, Jia B, Yan J, Zuniga-Hertz JP, Han C, Cai D. Hypothalamic stem cells control ageing speed partly through exosomal miRNAs. Nature. 2017 Aug 3;548(7665):52-57. doi: 10.1038/nature23282. Epub 2017 Jul 26. PMID 28746310
- [Background] Clegg A, Young J, Iliffe S, Rikkert MO, Rockwood K. Frailty in elderly people. Lancet. 2013 Mar 2;381(9868):752-62. doi: 10.1016/S0140-6736(12)62167-9. Epub 2013 Feb 8. PMID 23395245
- [Background] Song X, Mitnitski A, Rockwood K. Prevalence and 10-year outcomes of frailty in older adults in relation to deficit accumulation. J Am Geriatr Soc. 2010 Apr;58(4):681-7. doi: 10.1111/j.1532-5415.2010.02764.x. Epub 2010 Mar 22. PMID 20345864
- [Background] Lopez-Otin C, Blasco MA, Partridge L, Serrano M, Kroemer G. The hallmarks of aging. Cell. 2013 Jun 6;153(6):1194-217. doi: 10.1016/j.cell.2013.05.039. PMID 23746838
- [Background] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Background] Juma S, Taabazuing MM, Montero-Odasso M. Clinical Frailty Scale in an Acute Medicine Unit: a Simple Tool That Predicts Length of Stay. Can Geriatr J. 2016 Jun 29;19(2):34-9. doi: 10.5770/cgj.19.196. eCollection 2016 Jun. PMID 27403211
- [Background] Islam A, Muir-Hunter SW, Speechley M, Montero-Odasso M. Facilitating Frailty Identification: Comparison of Two Methods among Community-Dwelling Order Adults. J Frailty Aging. 2014;3(4):216-21. doi: 10.14283/jfa.2014.27. PMID 27048860